# UNIVERSITY OF WASHINGTON CONSENT FORM

# A Pilot Trial of 13-cis retinoic acid (Isotretinoin) for the Treatment of Men with Oligoasthenoteratozoospermia

# Researchers:

John K. Amory, MD, MPH, Professor, Medicine, 206-616-1727
Stephanie Page, MD, PhD, Associate Professor, Medicine, 206-616-0483
Mara Roth, MD, Assistant Professor, Medicine, 206-221-0519
Iris Nielsen, Research Coordinator, Medicine, 206-221-5473
Thomas Walsh, MD, Assistant Professor, Urology, 206-543-3640
Nina Isoherranen, PhD, Assistant Professor, Pharmaceutics, 206-543-2753
Charles Muller, PhD, Lecturer, Urology, 206-543-9504
William J. Bremner MD, PhD, Professor of Chairman, Medicine, 206-543-3293
Marilyn Buscher, RN, Medicine, 206-616-0482

This is the 24-hour emergency telephone number for the paging operator: 206-598-6190. Ask the operator to page one of these study doctors: Drs. Amory, Walsh, Page or Roth.

# Researchers' statement

We are asking you to be in a research study. The purpose of this consent form is to give you the information you will need to help you decide whether to be in the study or not. Please read the form carefully. You may ask questions about the purpose of the research, what we would ask you to do, the possible risks and benefits, your rights as a volunteer, and anything else about the research or this form that is not clear. When we have answered all your questions, you can decide if you want to be in the study or not. This process is called "informed consent." We will give you a copy of this form for your records.

#### PURPOSE OF THE STUDY

Our previous work has suggested that men with infertility may have low levels of the active form of Vitamin A, called retinoic acid, in their testes. We think that giving men with low sperm counts retinoic acid may increase their sperm counts and improve their chances of fathering a pregnancy. We are enrolling twenty men with infertility in a pilot research study here at the UW to see if retinoic acid administration over twenty weeks can increase sperm production and help infertile men become fathers. All men will receive retinoic acid treatment (there is no placebo group or blinding in this study).

#### STUDY PROCEDURES

This is a study to determine the impact of retinoic acid administration on sperm counts in men with infertility from low sperm counts.

To participate in the study you must be between 21-65 years of age and have infertility from a low sperm count, but be otherwise healthy. If you are currently taking anabolic steroids, illicit drugs or drink more than 4 alcoholic beverages daily, you cannot participate in this study. If you take medications such as lupron, ketoconazole, finasteride, dutasteride, methadone or lithium you cannot participate in this study.

The study involves 11 visits spaced out over 9-11 months.

All Study Visits will take place at the University of Washington

Screening 8-60 days – consists of two visits separated by one week.

# **Screening Visit 1 [Approximately 1 hour]**

Prior to any study procedures, you will be asked to read this informed consent form and ask any questions you may have. If you want to participate, you will then sign this consent form along with Dr. Amory. Next, Dr. Amory will review your medical history, ask you about the medications that you are taking and perform a physical examination, including measurement of your testicle size. A blood sample (about 2 tablespoons) will be drawn to assess your general health and measure the levels of hormones and vitamin A and retinoic acid levels in your blood, and you will be asked to complete a 9-question questionnaire about your mood. You may refuse to answer any question during this visit during the medical history or on the questionnaire. Finally, we will ask you to provide a sperm sample by masturbation after a minimum of 48 hours of no sexual activity to determine your sperm count, concentration, motility (movement) and morphology (appearance).

# **Screening Visit 2 (approximately 20 minutes)**

You will have a brief check of your blood pressure and pulse and be asked if you are taking any new medications. You will be asked to provide a 2<sup>nd</sup> baseline sperm sample after a minimum of 48 hours of no sexual activity

Treatment Visits. There are seven visits in the treatment period: week 0, 2, 4, 8, 12, 16, and 20. All visits are  $+\frac{4}{2}$  days. We will collect blood samples after 6 hours of fasting.

Treatment Visit 1 and 2, weeks 0 and 2 (approximately 45 minutes each)

This is the day 1 of treatment.

You will have a brief check of your blood pressure, pulse, and weight, and one of the study doctors will review how you are feeling and ask you about concomitant medications and adverse events. If you are taking a medication that is listed as disallowed you may be disallowed from the study. The doctor will perform a brief physical examination, including measurement of your testicle size. A blood sample (about 2 tablespoons) will be drawn to assess your general health and measure the levels of hormones and vitamin A and retinoic acid levels in your blood, and you will be asked to complete a 9-question questionnaire about your mood. You may refuse to answer any question during this visit during the medical history or on the questionnaire. We will also ask you to provide a sperm sample by masturbation after a minimum of 48 hours of no

sexual activity. Lastly, you will be given a 18-day supply of 13-cis retinoic acid (Isotretinoin) and a medication log and be instructed how to take and record your study drug use. We will ask that you not take study drug in the mornings of your visits, and bring unused study drug to each visit.

# Treatment Visits 3-6, (approximately 45 minutes each) weeks 4, 8, 12, and 16

You will have a brief check of your blood pressure and pulse and one of the study doctors will review how you are feeling and the presence of any new symptoms or possible side effects from the study medication and perform a brief physical examination, including measurement of your testicle size. A blood sample (about 2 tablespoons) will be drawn to assess your general health and measure the levels of hormones and vitamin A and retinoic acid levels in your blood, and you will be asked to complete a 9-question questionnaire about your mood. You may refuse to answer any question during this visit during the medical history or on the questionnaire. We will also ask you to provide a sperm sample by masturbation after a minimum of 48 hours of no sexual activity. Lastly, you will be given a 32-day supply of 13-cis retinoic acid (Isotretinoin) and a medication log.

# Treatment Visits 7, (approximately 45 minutes

You will have a brief check of your blood pressure and pulse and one of the study doctors will review how you are feeling and the presence of any new symptoms or possible side effects from the study medication and perform a brief physical examination, including measurement of your testicle size. A blood sample (about 2 tablespoons) will be drawn to assess your general health and measure the levels of hormones and vitamin A and retinoic acid levels in your blood, and you will be asked to complete a 9-question questionnaire about your mood. You may refuse to answer any question during this visit during the medical history or on the questionnaire. We will also ask you to provide a sperm sample by masturbation after a minimum of 48 hours of no sexual activity.

# Follow-up Visits 1 and 2 (45 minutes each), weeks 24 and 32, $\pm$ 4 days

You will have a brief check of your blood pressure and pulse and one of the study doctors will review how you are feeling and the presence of any new symptoms and perform a brief physical examination, including measurement of your testicle size. A blood sample (about 2 tablespoons) will be drawn to assess your general health and measure the levels of hormones and vitamin A and retinoic acid levels in your blood, and you will be asked to complete a 9-question questionnaire about your mood. You may refuse to answer any question during this visit during the medical history or on the questionnaire. We will also ask you to provide a sperm sample by masturbation after a minimum of 48 hours of no sexual activity.

#### RISKS, STRESS, OR DISCOMFORT

**Medical History:** The interview with the study doctor and medical form includes questions about your medical history, which may cause you some discomfort or embarrassment. You are free to refuse to answer any of these questions.

**Blood draws**: Blood draws can cause some discomfort and occasionally lightheadedness, or fainting in some subjects. There is also a risk of infection or bruising around the sight of the blood draw. A bruise may form where the needle enters the vein.

**Laboratory results:** We will share all of your test results with you, including any changes in your sperm counts. If any of your lab results are abnormal, we may have you return for a repeat blood draw. If any of the results are abnormal, especially if it is worrisome in terms of your health or means you cannot participate in the study, we will let you know immediately.

**Confidentiality:** As indicated in the section below, your identity will be kept confidential. However, in the very unlikely event of a breach of confidentiality, there is a risk you would experience a feeling of invasion of your privacy.

**Medications:** 13-cis retinoic acid therapy (Isotretinoin) is commonly used for the treatment of severe acne. It can be associated with significant side effects including tiredness (10%), eczema of the skin or inflammation of the lips (15%) and rarely depression (<1%). If these side effects become severe, it may be necessary to stop drug administration. If you experience study-related injury, illness, or distress, please contact Dr. Amory, Page, Roth or Walsh at the numbers above immediately.

Because 13-cis retinoic acid (Isotretinoin) treatment for infertility is experimental, it is unknown if treatment will improve your sperm counts. Please know that we will provide you with any information developed during the study that might affect your willingness to participate.

#### ALTERNATIVES TO TAKING PART IN THIS STUDY

You are participating in this study as a man with infertility due to a reduced sperm count. The alternative to participation is not to participate and use IVF or donor sperm to treat your infertility.

# BENEFITS OF THE STUDY

Information from this study may be useful in the treatment of men with infertility from low sperm counts.

# MEDICAL RECORD INFORMATION

Policies require that we put information about this research into your permanent medical record at UW Medicine. If you do not have a medical record at UW Medicine, one will be created for you even if your only connection with UW Medicine is as a research subject.

# Information that will be put into your medical record:

1. Your name, address, telephone number, date of birth, social security number, health insurance information, billing information, and any other information you provide on the hospital or clinic information form.

# 2. Information about this research study:

- Name of the study, described as: [RRRRA, TWO]
- The name of the researcher
- The name of the study coordinator
- Contact phone number for the study
- Contact email address for the study
- Emergency phone number for the study
- Expected start and end dates for your time in the study

#### Who will have access

This medical record will be permanent. It will be stored with all other UW Medicine medical records. A copy of your record may also be stored on the secure UW Medicine medical record computer system. Access to medical records and the computer system is restricted to only authorized staff with passwords for the system. Only UW Medicine staff and people who have legal access to your medical record will be able to see it. This may include your insurance company and government regulatory agencies. If you have already given permission to anyone (such as your health insurance company) to look at your medical record, they may receive this research information if they ask for a copy of your medical record.

#### Your health insurance

Though very unlikely, this could have some effect on what your health insurance company (but not Medicaid or Medicare) is willing to pay for while you are in the research. If this infrequent situation happens, we may be able to help by giving you some information to share with your health insurance company.

#### **SOURCE OF FUNDING**

The study team and/or the University of Washington is receiving grant funding for this research from the Eunice Kennedy Shriver National Institute of Childhood Health and Human Development, the part of the National Institutes of Health that performs infertility research.

#### CONFIDENTIALITY OF RESEARCH INFORMATION

Your lab results and sperm count data will be kept in a private research chart in the lab, and will not be placed in your medical record.

All study data will be confidential with a link between your data and your assigned study number. This link will be retained until 1/1/2020 after which point your data will be made anonymous.

All of the information you provide will be confidential. However, if we learn that you intend to harm yourself or others, we must report that to the authorities.

Government or university staff sometimes review studies such as this one to make sure they are being done safely and legally. If a review of this study takes place, your records may be examined. The reviewers will protect your privacy. The study records will not be used to put you at legal risk of harm.

The U.S. Food and Drug Administration (FDA) reserves the right to review study data that may contain identifying information.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### OTHER INFORMATION

All study treatment procedures will be provided at no cost to you throughout your participation in this study. You will receive up to \$390 for completion of this study to cover the costs of your time, travel, and inconvenience. You will receive \$30 after the 1<sup>st</sup> screening and \$20 after the 2<sup>nd</sup> screening visit. You will receive \$40 for each study visit during the treatment phase and \$30 for each of the two follow-up visits. If we request that you return to repeat a screening lab test, you will receive an additional \$25 for your time and inconvenience. In addition we will provide you with parking validation or a metro transit token. If you are not a citizen of the United States and do not have a social security number, we are required to withhold 30% of your payment for taxes.

The researchers will keep the link between your name and study number for up to six years, which means they will destroy the link no later than January 1<sup>st</sup>, 2020. We will keep your blood samples, labeled with your study identification number and initials for 5 years after the end of the study. After that point, we will remove all identifying information from your blood samples. We keep these samples in the event that more effective ways for understanding the relationship between retinoic acid and sperm production become available.

By signing this consent form, you agree to allow the researchers to decide what to do with any surplus samples (blood and semen) removed from your body during the research described above. No sperm will be used to fertilize an egg for research purposes. You will be told if the researcher has any current personal interest, such as any economic interest, related to performing this research (there is none). The semen samples will be stored for future analysis as well for up to six years to understand the presence of Isotretinoin in the semen. The serum samples may be used for the assessment of newly developed hormone assays or bioassays when available. You may contact the investigator to discard your samples after the aims of the study have been met, no sooner than five years after the study closes.

You must inform your study doctor of any drugs you use during the study and of any illness that develops (of any type or severity) while participating in this study.

Your taking part in this study may be stopped at any time. The study doctor can stop the study without your consent for the following reasons:

- it appears to be medically harmful to you;
- missing scheduled clinic visits;

- refusal to complete required tests;
- development of a medical condition(s) or serious side effect(s) that may pose a health risk to you;
- you do not meet the study requirements;
- the study is cancelled;
- for administrative reasons including enrollment (the target number of subjects have been enrolled) or
- for any other reason

Your participation is voluntary. You may refuse to participate and are free to withdraw from this study at any time without penalty or loss of benefits to which you are otherwise entitled. If you do withdraw, however, we will ask you to return to the clinic for any study tests necessary in insure your safety and well-being. Your decision will not adversely affect your medical care.

#### **COMPENSATION FOR INJURY**

In the event that physical illness or injury occurs as a direct result of study procedures, contact the study staff [Dr. Amory, (206) 616-1727] right away. The study staff will treat you or refer you for treatment. The UW will pay up to \$10,000 to treat injury or illness caused by the study. No money has been set aside to pay for things like lost wages, lost time, or pain. However, you will not lose your legal right to seek payment if you sign this form.

| Printed name of study staff obt | aining consent | Signature | Date | |
|---|---|---|---|---|
| Subject's statement | | | | |
| This study has been explained to chance to ask questions. If I have researchers listed above. If I have Human Subjects Division at (2) | ave questions later<br>ave questions abou | about the reseaut my rights as a | rch, I can ask<br>a research sub | one of the pject, I can call the |
| Printed name of subject | Signature o | f subject | | Date |
| Copies to: Researcher | | | | |

Subject

Subject's Medical Record (if applicable)

# **Appendix 1: Schedule of Events**

| | | Screening | | Treatment (± 4 days) | | Follow-up (± 4 days) | |
|---|---|---|---|---|---|---|---|
| | Visit # | S1 | S2 | T1 | T2-T7 | F1 | F2 |
| | Study Day | -60 to -1 | -53 to 1 | 1 | Wks: 2, 4, 8, 12, 16, 20 | Wk 24 | Wk 32 |
| Administrative | Informed consent/HIPAA | X | | | | | |
| | Vital Signs | X | X | X | X | X | X |
| Medical | Medical History | X | | | | | |
| | Physical Exam | X | | X | X | X | X |
| - | AE & Con Med | X | X | X | X | X | X |
| | Semen Analysis | X | X | X | X | X | X |
| | PHQ9<br>Questionnaire | X | | X | X | X | X |
| Blood Sampling | CBC, Chemistry,<br>Lipids, CK | X | | X | X | X | X |
| | FSH, LH, T &<br>Retinoids | X | | X | X | X | X |
| Administration M Di m Cc re Cc | Dispense Study<br>Meds | | | X | X | | |
| | Dispense study med log | | | X | X | | |
| | Collect and review med log | | | | X | | |
| | Collect unused study meds | | | | X | | |
| Reimbursement (\$) | | 30 | 20 | 40 | 40 | 30 | 30 |

# **Abbreviations:**

HIPAA: Health insurance portability and accountability act

PHQ9: Patient health questionnaire, #9 FSH: follicle-stimulating hormone

LH: luteinizing hormone

T: testosterone AE: adverse event

Con Med: concomitant medications

S1/S2: screening visit 1/2 T1-T7: treatment visits 1-7 F1/F2: follow-up visit 1/2

Wk: week